CLINICAL TRIAL: NCT05650112
Title: A Study of the Safety, Tolerability, Microbial Kinetics and Effect on Urinary Oxalate Excretion of FB-001 in Healthy Volunteers Fed a High Oxalate/Low Calcium Diet and in Patients With Enteric Hyperoxaluria
Brief Title: Safety and Tolerability of FB-001 in Healthy Adult Volunteers and Adult Subjects With Enteric Hyperoxaluria
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federation Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FB-001-101
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Healthy; Enteric Hyperoxaluria
Keywords: Enteric Hyperoxaluria; Gastrointestinal disorder; Fat malabsorption; Urinary oxalate; Kidney stones; Live Biotherapeutic Product
MeSH Terms: conditions — Gastrointestinal Diseases; Kidney Calculi

STUDY DESIGN:
Intervention Model Description: Part 1 - randomized, placebo-controlled. Part 2 - open label.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Part 1 is double blind. Part 2 is open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- FB-001 Healthy Volunteer (Experimental): Healthy volunteer participants in Part 1 receive FB-001 (1 x 10^12 viable cells) orally on Day 1 and Day 2 and FB-001 (1 x 10^11 viable cells) orally on Days 3 to 10.
  Interventions: Biological: FB-001
- Placebo (Placebo Comparator): Healthy volunteer participants receive placebo once a day, orally, for 10 days in Part 1.
  Interventions: Biological: Placebo
- FB-001 Enteric Hyperoxaluria (Experimental): Enteric hyperoxaluria participants in Part 2 receive FB-001 (1 x 10^12 viable cells) orally on Day 1 and Day 2 and FB-001 (1 x 10^11 viable cells) orally on Days 3 to 10.
  Interventions: Biological: FB-001

INTERVENTIONS:
Biological: FB-001 — FB-001 is formulated as a powder in capsule intended for oral administration
  Arms: FB-001 Enteric Hyperoxaluria; FB-001 Healthy Volunteer
Biological: Placebo — In order to maintain study blinding, matching placebo in identical packaging is manufactured using an inactive powder in capsule
  Arms: Placebo

SUMMARY:
This Phase 1, first-in-human, randomized, double-blinded, placebo controlled study is evaluating FB-001 in healthy volunteers (Part 1) and participants diagnosed with enteric hyperoxaluria (Part 2). Eligible participants receive investigational product and undergo safety monitoring, evaluations and subsequent follow-up after investigational product administration.

DETAILED DESCRIPTION:
This study is evaluating the safety, tolerability and microbial kinetics of FB-001 within the following 2 study parts:

Part 1 is an inpatient, placebo-controlled, study in 32 healthy volunteer male and female participants (16 treated: 16 placebo) for 10 days of dosing consisting of a loading dose of 1 × 10^12 viable cells administered orally on Day 1 and Day 2 and a dose of 1 × 10^11 viable cells administered orally on Day 3 to Day 10.

Part 2 is an outpatient open label study in up to 16 adult male and female participants with enteric hyperoxaluria, defined as increased gastrointestinal oxalate absorption in the context of fat malabsorption and/or increased intestinal permeability to oxalate caused by gastrointestinal disorders. Participants will receive FB-001 for 10 days consisting of a loading dose of 1 × 10^12 viable cells administered orally on Day 1 and Day 2 and a dose of 1 × 10^11 viable cells administered orally on Day 3 to Day 10.

ELIGIBILITY:
Part 1 Key Inclusion Criteria:

1. ≥ 18 to ≤ 50 years.
2. Willing to participate and sign the informed consent form.
3. Available for and agree to comply with all study requirements, including duration of stay at the clinical pharmacology unit, adherence to diet control, study drug administration, follow-up visits, and collection of stool, urine, and blood.
4. Normal clinical laboratory test results which are not considered to be clinically significant by the Investigator at Screening (including an estimated glomerular filtration rate [eGFR] >60 mL/min/1.73 m2 calculated using the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] equation).
5. Body mass index (BMI) 18 to 35 kg/m2.
6. Volunteers must have 24-hour urinary oxalate <45 mg.

Part 1 Key Exclusion Criteria:

1. Presence or history of any significant cardiovascular, gastrointestinal, hepatic, renal, pulmonary, hematologic, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease, as determined by the Investigator.
2. Presence or history of any condition or procedure (including surgery) known to interfere with the absorption, distribution, metabolism, or excretion of medicines.
3. Participation in any study of an investigational product, biologic, device, or other agent within 30 days prior to admission on Day -7 or unwilling to forego other forms of investigational treatment during this study.
4. Major surgery or an inpatient hospital stay within 3 months prior to admission on Day -7.
5. A positive serologic test for infection with human immunodeficiency virus, hepatitis C virus, or hepatitis B virus.
6. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin >1.5 × upper limit of normal (ULN).
7. Hemoglobin A1c (HbA1c) ≥6.5 percent.
8. Hyperthyroidism or hypothyroidism as defined by thyroid-stimulating hormone (TSH) levels outside the normal reference range.
9. History of QT prolongation or dysrhythmia or a family history of prolonged QT interval or sudden death.
10. Use of prescription drugs (except for hormonal contraceptives) including cisapride, pimozide, astemizole, terfenadine, ergotamine, or dihydroergotamine within 4 weeks prior to Screening and unable or unwilling to refrain from such use through the end of study visit.
11. Use of any herbal or over-the-counter medications, probiotic products, or vitamin supplements, including vitamin C, within 14 days prior to first administration of study drug through the end of the Confinement Period.
12. Planned procedures that may require antibiotics between Screening and the end of study visit.
13. Use of antibiotic treatment up to 4 weeks prior to or during Screening, or between Screening and admission (Day -7), or a history of recurrent infections requiring antibiotics.
14. A known hypersensitivity to MiraLax, clarithromycin, erythromycin, any of the macrolide antibiotics, metronidazole or other nitroimidazole derivatives.
15. A history of kidney stones.
16. Unwilling to comply with all study procedures and assessments, including the High Oxalate Low Calcium (HOLC) diet and the pretreatment regimen, which includes antibiotics.

Part 2 Key Inclusion Criteria:

1. ≥ 18 to ≤ 74 years.
2. Willing to participate and sign the informed consent form.
3. Available for and agree to comply with all study requirements, including study drug administration, follow-up visits, and collection of stool, urine, and blood.
4. Body Mass Index (BMI) 18 to 40 kg/m2.
5. Enteric hyperoxaluria diagnosis as indicated by 24-hour urinary oxalate levels of ≥50 mg at Screening. Enteric hyperoxaluria is defined as increased gastrointestinal oxalate absorption in the context of fat malabsorption and/or increased intestinal permeability to oxalate caused by gastrointestinal disorders.
6. Screening laboratory evaluations (eg, chemistry panel, complete blood count with differential, prothrombin time/activated partial thromboplastin time, urinalysis) and a 12-lead ECG that are within normal limits or judged to be not clinically significant by the Investigator.
7. Patients on concomitant medication for management of kidney stone risk factors (eg, calcium supplements, thiazide diuretics, allopurinol, and alkali therapy) must be on stable dose regimen for at least 8 weeks prior to Screening, with no changes in dosing (dose level or dosing frequency) anticipated during the study Treatment Period.

Part 2 Key Exclusion Criteria:

1. Presence or history of any significant cardiovascular, gastrointestinal, hepatic, renal, pulmonary, hematologic, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease, as determined by the Investigator.
2. Presence or history of any condition or procedure (including surgery) known to interfere with the absorption, distribution, metabolism, or excretion of medicines.
3. Participation in any study of an investigational product, biologic, device, or other agent within 30 days prior to Visit 1 (Day -7) or are not willing to forego other forms of investigational treatment during this study.
4. Major surgery or an inpatient hospital stay within 3 months prior to Visit 1 (Day -7).
5. Uncontrolled hypertension with systolic blood pressure >160 mmHg and diastolic blood pressure >100 mmHg.
6. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2 × upper limit of normal (ULN) or total bilirubin >1 × ULN at Screening unless the patient has known Gilbert's syndrome.
7. Hemoglobin A1c (HbA1c) ≥6.5 percent.
8. Hyperthyroidism or hypothyroidism as defined by thyroid stimulating hormone (TSH) levels outside the normal reference range.
9. History of QT prolongation or dysrhythmia, or a family history of prolonged QT interval or sudden death.
10. Estimated glomerular filtration rate (eGFR) <45 mL/min/1.73 m2 calculated using the CKD-EPI equation.
11. Loose or liquid stools (Bristol Stool Scale Type 6 or 7) within 1 week prior to or during Screening.
12. Consumption of any herbal medications, probiotic products, or vitamin supplements, including vitamin C, within 14 days prior to first administration of study drug through the end of the Treatment Period.
13. Chronic therapy with high doses of systemic steroids (>10 mg/day prednisone or equivalent daily) or intensification of existing immunosuppressant or immunomodulatory therapy for treatment of an acute disease flare within 4 weeks prior to or during Screening.
14. Planned procedures that may require antibiotics between Screening and the end of study visit.
15. Use of antibiotic treatment up to 4 weeks prior to or during Screening, or between Screening and Visit 1 (Day -7), or a history of recurrent infections requiring antibiotics.
16. A known hypersensitivity to MiraLax, clarithromycin, erythromycin, any of the macrolide antibiotics, metronidazole, or other nitroimidazole derivatives.
17. Unable or unwilling to discontinue use of cisapride, pimozide, astemizole, terfenadine, ergotamine, or dihydroergotamine from Visit 1 (Day -7) through the end of study visit.
18. A known genetic, congenital, or other known causes of kidney stones (eg, primary hyperoxaluria, cystinuria, primary hyperparathyroidism, or medullary sponge kidney).
19. A history of Roux-en-Y gastric bypass or other bariatric surgery procedures within 6 months prior to Screening.
20. Inflammatory bowel disease that is clinically unstable or have a change in medication to control disease activity within 4 weeks prior to Screening.
21. Unwilling to comply with all study procedures and assessments, including need for pretreatment regimen which includes antibiotics.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-11-16 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects With Treatment-Emergent Adverse Events | 196 days
  Toxicity is graded in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0. Adverse events (AEs) are reported based on clinical laboratory tests, vital signs, physical examinations, electrocardiograms, and any other medically indicated assessments from the time informed consent is signed through the end of the safety follow-up period. AEs are considered to be treatment emergent (TEAE) if they occur or worsen in severity after the first dose of study treatment. TEAEs are considered treatment-related if relationship to study drug is possibly related, probably related, or definitely related.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Grauer, MD, Study Director — Chief Medical Officer
Locations (1):
- Medpace Clinical Pharmacology Unit, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No